CLINICAL TRIAL: NCT02476279
Title: Stent vs. Indomethacin for Preventing Post-ERCP Pancreatitis: The SVI Trial
Brief Title: Stent vs. Indomethacin for Preventing Post-ERCP Pancreatitis
Acronym: SVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Badih Joseph Elmunzer, Professor of Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01DK104833-01 (NIH); U01DK104833-01 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Results first posted 2024-05-08 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-04

CONDITIONS: Post-ERCP Pancreatitis
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin alone (Experimental): Indomethacin 100 mg rectally immediately after ERCP
  Interventions: Other: Indomethacin 100 mg rectally immediately after ERCP, NO prophylactic pancreatic stent placement
- Indomethacin+pancreatic stent (Active Comparator): Indomethacin 100 mg rectally immediately after ERCP AND prophylactic pancreatic stent placement
  Interventions: Other: Indomethacin 100 mg rectally immediately after ERCP AND prophylactic pancreatic stent placement

INTERVENTIONS:
Other: Indomethacin 100 mg rectally immediately after ERCP, NO prophylactic pancreatic stent placement
  Arms: Indomethacin alone
Other: Indomethacin 100 mg rectally immediately after ERCP AND prophylactic pancreatic stent placement
  Arms: Indomethacin+pancreatic stent

SUMMARY:
Background: Pancreatitis is the most frequent complication of endoscopic retrograde cholangiopancreatography (ERCP), accounting for substantial morbidity, occasional mortality, and increased health care expenditures. Until recently, the only effective method of preventing post-ERCP pancreatitis (PEP) had been prophylactic pancreatic stent placement (PSP), an intervention that is costly, time consuming, technically challenging, and potentially dangerous. The investigators recently reported the results of a large randomized controlled trial demonstrating that rectal indomethacin, a non-steroidal anti-inflammatory drug, reduced the risk of pancreatitis after ERCP in high-risk patients, most of whom (>80%) had received a pancreatic stent. Secondary analysis of this RCT suggested that subjects who received indomethacin alone were less likely to develop PEP than those who received a pancreatic stent alone or the combination of indomethacin and stent, even after adjusting for underlying differences in subject risk. If indomethacin were to obviate the need for PSP, major clinical and cost benefits in ERCP practice could be realized.

Objective: To assess whether rectal indomethacin alone is non-inferior to the combination of rectal indomethacin and prophylactic pancreatic stent placement for preventing post-ERCP pancreatitis in high-risk cases.

Methods: Comparative effectiveness multi-center non-inferiority trial of rectal indomethacin alone vs. the combination of rectal indomethacin and prophylactic pancreatic stent placement for the prevention of post-ERCP pancreatitis in high-risk patients. One thousand four hundred and thirty subjects at elevated risk for PEP who would normally receive a pancreatic stent for prophylaxis will be randomized to indomethacin alone or the combination of indomethacin and PSP. The proportion of patients developing PEP and moderate-severe PEP will be compared. In addition, the investigators will establish a quality-assured central repository of biological specimens obtained from study participants, permitting future translational research elucidating the molecular and genetic mechanisms of PEP, as well as the mechanisms by which non-steroidal anti-inflammatory drugs prevent this complication.

DETAILED DESCRIPTION:
The purpose of the SVI study is to determine whether or not rectal indomethacin has no important loss of efficacy as compared to the combination of rectal indomethacin and prophylactic pancreatic stent placement in patients undergoing high-risk ERCP who require pancreatic stent placement (PSP) for the sole purpose of pancreatitis prevention. The primary efficacy endpoint is defined as post-ERCP pancreatitis defined per consensus (Altanta) criteria. Another way of stating the trial's purpose is that the proportion of subjects with post-ERCP pancreatitis on rectal indomethacin alone is not more than that of the combination of rectal indomethacin and prophylactic PSP by more than a pre-specified absolute amount (i.e., the non-inferiority margin).

This is a blinded, two-armed non-inferiority trial where eligible patients will be randomized to either the combination treatment or indomethacin alone. Participants will be randomized during the ERCP procedure after eligibility is confirmed, and receive indomethacin at the time of randomization. The primary efficacy endpoint of post-ERCP pancreatitis within 2 days from randomization will be assessed by an independent adjudication panel. The participant follow-up period is 30 days from randomization.

ELIGIBILITY:
Inclusion Criteria:

Any patient undergoing ERCP in whom pancreatic stent placement is planned for post-ERCP pancreatitis prevention, is ≥ 18 years old, who provides informed consent, AND:

Has one of the following:

1. Clinical suspicion of or known sphincter of Oddi dysfunction
2. History of post-ERCP pancreatitis (at least one prior episode of pancreatitis after ERCP)
3. Pancreatic sphincterotomy
4. Pre-cut (access) sphincterotomy (freehand pre-cut and septotomy)
5. Difficult cannulation: cannulation duration ≥ 6 minutes (starting at time of initial papillary engagement with at least 25% of the time in contact with the papilla) AND/OR ≥ 6 cannulation attempts (defined as sustained contact with papilla lasting at least 1 second).
6. Short-duration (≤ 1 min) balloon dilation of an intact biliary sphincter.

   Or has at least 2 of the following:
7. Age < 50 years old & female gender
8. History of recurrent pancreatitis (at least 2 episodes)
9. ≥3 pancreatic injections
10. Pancreatic acinarization
11. Pancreatic brush cytology

Exclusion Criteria:

1. Ampullectomy
2. Cases in which a pancreatic stent must be placed for therapeutic intent
3. Unwillingness or inability to consent for the study
4. Pregnancy
5. Breast feeding mother
6. Standard contraindications to ERCP
7. Allergy to Aspirin or NSAIDs
8. Known renal failure (Cr > 1.4 mg/dl)
9. Ongoing or recent (within 2 weeks) hospitalization for gastrointestinal hemorrhage
10. Ongoing or recent (within 1 week) hospitalization for acute pancreatitis
11. Known chronic calcific pancreatitis
12. Pancreatic head malignancy
13. Procedure performed on major papilla/ventral pancreatic duct in patient with pancreas divisum (no manipulation of minor papilla)
14. ERCP for biliary stent removal or exchange without anticipated pancreatogram
15. Subjects with prior biliary sphincterotomy now scheduled for repeat biliary therapy without anticipated pancreatogram
16. Anticipated inability to follow protocol
17. Absence of rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1950 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Univesrity of Southern California, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - The Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Dartmouth University, Lebanon, New Hampshire
  - Case Western Reserve University, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Calgary, Calgary
  - McGill University, Montreal

REFERENCES:
- [Derived] Elmunzer BJ, Foster LD, Serrano J, Cote GA, Edmundowicz SA, Wani S, Shah R, Bang JY, Varadarajulu S, Singh VK, Khashab M, Kwon RS, Scheiman JM, Willingham FF, Keilin SA, Papachristou GI, Chak A, Slivka A, Mullady D, Kushnir V, Buxbaum J, Keswani R, Gardner TB, Forbes N, Rastogi A, Ross A, Law J, Yachimski P, Chen YI, Barkun A, Smith ZL, Petersen B, Wang AY, Saltzman JR, Spitzer RL, Ordiah C, Spino C, Durkalski-Mauldin V; SVI Study Group. Indomethacin with or without prophylactic pancreatic stent placement to prevent pancreatitis after ERCP: a randomised non-inferiority trial. Lancet. 2024 Feb 3;403(10425):450-458. doi: 10.1016/S0140-6736(23)02356-5. Epub 2024 Jan 11. PMID 38219767
- [Derived] Elmunzer BJ, Serrano J, Chak A, Edmundowicz SA, Papachristou GI, Scheiman JM, Singh VK, Varadarajulu S, Vargo JJ, Willingham FF, Baron TH, Cote GA, Romagnuolo J, Wood-Williams A, Depue EK, Spitzer RL, Spino C, Foster LD, Durkalski V; SVI study group and the United States Cooperative for Outcomes Research in Endoscopy (USCORE). Rectal indomethacin alone versus indomethacin and prophylactic pancreatic stent placement for preventing pancreatitis after ERCP: study protocol for a randomized controlled trial. Trials. 2016 Mar 3;17(1):120. doi: 10.1186/s13063-016-1251-2. PMID 26941086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 20 referral centers in the USA and Canada between September 2015 and January 2023.
Pre-assignment Details: Of 7243 patients assessed for eligibility, 1950 met eligibility criteria and were randomly assigned to treatment.
Groups:
- Indomethacin Alone: Indomethacin 100 mg rectally immediately after ERCP, NO prophylactic pancreatic stent placement
Period: Overall Study
Arm/Group | Indomethacin Alone | Indomethacin+Pancreatic Stent
Started | 975 | 975
Completed (Completed follow-up for the primary and secondary endpoints) | 974 | 974
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin Alone | Indomethacin+Pancreatic Stent | Total
Number analyzed (Participants) | 975 | 975 | 1950
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (16.4) | 55.8 (16.3) | 55.7 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 599 | 596 | 1195
  Male | 376 | 379 | 755
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 99 | 200
  Not Hispanic or Latino | 866 | 871 | 1737
  Unknown or Not Reported | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 115 | 102 | 217
  White | 809 | 825 | 1634
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 26 | 17 | 43
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI missing for 3 participants
  kg/m^2
    number analyzed (Participants) | 972 | 975 | 1947
    (all) | 28.6 (6.8) | 29.6 (7.2) | 29.1 (7.0)
Antibiotic use in past 3 months [Count of Participants; unit: Participants] — Population: Missing in 207 patients (100 in indomethacin plus stent group, 107 in indomethacin alone group) due to question being added in August, 2016.
  Participants
    number analyzed (Participants) | 868 | 875 | 1743
    (all) | 363 | 366 | 729
Clinical suspicion or known sphincter of Oddi dysfunction [Count of Participants; unit: Participants] | 262 | 252 | 514
History of post-ERCP pancreatitis [Count of Participants; unit: Participants] | 36 | 24 | 60
History of recurrent pancreatitis [Count of Participants; unit: Participants] | 128 | 126 | 254
Difficult cannulation [Count of Participants; unit: Participants] | 795 | 823 | 1618
Precut (access) sphincterotomy [Count of Participants; unit: Participants] | 112 | 100 | 212
Number of pancreatic injections [Median (Inter-Quartile Range); unit: injections] — Population: Missing in three patients (one in indomethacin plus stent group, two in indomethacin alone group).
  injections
    number analyzed (Participants) | 973 | 974 | 1947
    (all) | 0 [0 to 1] | 1 [0 to 2] | 1 [0 to 2]
Pancreatic sphincterotomy [Count of Participants; unit: Participants] | 58 | 66 | 124
Pancreatic acinarisation [Count of Participants; unit: Participants] | 6 | 8 | 14
Biliary sphincterotomy [Count of Participants; unit: Participants] | 864 | 869 | 1733
Trainee involvement [Count of Participants; unit: Participants] — All ERCPs were performed or directly supervised by board certified gastroenterologists with specialized expertise in ERCP who are faculty physicians at participating study centers. Some ERCPs involved trainees at varying stages of ERCP proficiency.
  Participants | 555 | 546 | 1101
Total intravenous fluid received during periprocedural period, mL [Mean (Standard Deviation); unit: mL] — Population: Missing in two patients (one in indomethacin plus stent group, one in indomethacin alone group).
  mL
    number analyzed (Participants) | 974 | 974 | 1948
    (all) | 1796 (935) | 1852 (938) | 1824 (937)
Total intravenous lactated Ringer's fluid received during periprocedural period, mL [Mean (Standard Deviation); unit: mL] — Population: Missing in five patients (two in indomethacin plus stent group, three in indomethacin alone group).
  mL
    number analyzed (Participants) | 972 | 973 | 1945
    (all) | 1554 (1052) | 1606 (1085) | 1581 (1069)
Prophylactic pancreatic stent calibre in those who received a stent [Count of Participants; unit: Participants] — Population: Analysis population is those who received a stent. Participants that received a stent in the Indomethacin Alone arm and participants that did not receive a stent in the Indomethacin+ Pancreatic Stent arm are treatment crossovers.
  Participants
    number analyzed (Participants) | 16 | 787 | 803
    3 French | 0 | 18 | 18
    4 French | 4 | 165 | 169
    5 French | 9 | 586 | 595
    >5 French | 0 | 18 | 18
    Missing | 3 | 0 | 3
Prophylactic pancreatic stent length in those who received a stent [Count of Participants; unit: Participants] — Population: Analysis population is those who received a stent. Participants that received a stent in the Indomethacin Alone arm and participants that did not receive a stent in the Indomethacin+ Pancreatic Stent arm are treatment crossovers.
  Participants
    number analyzed (Participants) | 16 | 787 | 803
    2-5cm | 7 | 455 | 462
    6-8cm | 3 | 95 | 98
    >8cm | 3 | 237 | 240
    Missing | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects in Each Study Group With Post-ERCP Pancreatitis
Description: Post-ERCP pancreatitis (PEP) was based on a widely validated consensus definition that was applied as a diagnostic framework. In this consensus definition, PEP is diagnosed if there was new onset (or increase) of pain in the upper abdomen, elevation in pancreatic enzymes of at least three times the upper limit of normal 24 h after the procedure, and hospitalization for at least two nights. The outcome was independently adjudicated by 3 ERCP experts at non-enrolling centers based on review of the medical records for study participants who were hospitalized with any adverse event within 2 days of the ERCP. Medical records were redacted of all information that could potentially reveal study group assignment, including radiology reports. The consensus definition was applied as a diagnostic framework so that adjudicators could use their best judgment in cases that did not strictly satisfy the criteria. PEP was declared if there was agreement between at least two of the three adjudicators.
Time Frame: Within 48 hours after ERCP
Population: Intention-To-Treat and Per Protocol populations
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin Alone | Indomethacin+Pancreatic Stent
Number analyzed (Participants) | 975 | 975
Participants
  Intention-To-Treat Population | 145 | 110
  Per Protocol Population: number analyzed (Participants) | 951 | 777
  Per Protocol Population | 137 | 90
Statistical Analysis 1: Comparison: Indomethacin Alone vs Indomethacin+Pancreatic Stent; Test type: Non-Inferiority — To declare noninferiority, the upper bound of the two-sided 95% CI for the risk difference in post-ERCP pancreatitis (indomethacin alone minus indomethacin plus stent) needed to be less than 5% in both the intention-to-treat and per protocol analysis populations; Risk Difference (RD) = 0.036, 95% CI 2-sided [0.006 to 0.066] — These numbers are in the intention-to-treat analysis population. Risk difference in post-ERCP pancreatitis (PEP) is calculated as risk of PEP in indomethacin alone arm minus risk of PEP in indomethacin plus stent arm
Statistical Analysis 2: Comparison: Indomethacin Alone vs Indomethacin+Pancreatic Stent; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.003 to 0.060] — These numbers are in the per protocol analysis population. Risk difference in post-ERCP pancreatitis (PEP) is calculated as risk of PEP in indomethacin alone arm minus risk of PEP in indomethacin plus stent arm

2. Secondary Outcome: The Proportion of Subjects in Each Study Group With Moderate-severe Post-ERCP Pancreatitis
Description: Moderate or severe post-ERCP pancreatitis was based on the consensus definition as a diagnostic framework. For the severity assessment, radiographic information was made available to the adjudicators. The severity was defined as mild post-ERCP pancreatitis resulting in a hospitalization of ≤3 days, moderate post-ERCP pancreatitis resulting in a hospitalization of 4-10 days, and severe post-ERCP pancreatitis resulting in a hospitalization of > 10 days, or leading to the development of pancreatic necrosis or pseudocyst, or requiring percutaneous or surgical intervention. The outcome was declared if there was agreement between at least two of the three adjudicators.
Time Frame: Within one month of ERCP
Population: Intention-to-treat and per protocol. Outcome data missing for two participants (one in each treatment arm) and excluded from percentage denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin Alone | Indomethacin+Pancreatic Stent
Number analyzed (Participants) | 974 | 974
Participants
  Intention-to-treat population | 78 | 58
  Per protocol population: number analyzed (Participants) | 951 | 777
  Per protocol population | 74 | 45
Statistical Analysis 1: Comparison: Indomethacin Alone vs Indomethacin+Pancreatic Stent; Test type: Other; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.002 to 0.043] — These numbers are in the intention-to-treat analysis population. Risk difference is calculated as risk of moderate-severe PEP in indomethacin alone arm minus risk of moderate-severe PEP in indomethacin plus stent arm
Statistical Analysis 2: Comparison: Indomethacin Alone vs Indomethacin+Pancreatic Stent; Test type: Other; Risk Difference (RD) = 0.020, 95% CI 2-sided [-0.004 to 0.044] — These numbers are in the per protocol analysis population. Risk difference is calculated as risk of moderate-severe PEP in indomethacin alone arm minus risk of moderate-severe PEP in indomethacin plus stent arm

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected from randomization through the Day 5 follow up visit. Serious adverse events were collected from randomization through the end of study (Day 30).
Description: Adverse events were assessed at two follow up visits post-randomization: (1) 3-5 days after ERCP and (2) 30 (+/-5) days after ERCP. The follow-up was accomplished by directly contacting the subject or their treating healthcare provider in the event he or she had been hospitalized.
Arm/Group | Indomethacin Alone | Indomethacin+Pancreatic Stent
All-Cause Mortality (participants affected / at risk) | 24/975 | 26/975
Serious Adverse Events (participants affected / at risk) | 355/975 | 352/975
Other Adverse Events (participants affected / at risk) | 233/975 | 228/975
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin Alone (N=975) | Indomethacin+Pancreatic Stent (N=975)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 140 (163) | 166 (177)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 8 (8)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 2 (2)
Haemorrhagic necrotic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 9 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 16 (16) | 9 (9)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 90 (92) | 76 (80)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Perforation (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 6 (6)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 11 (11) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 4 (6)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (2) | 3 (3)
Biliary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder abscess (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 10 (10) | 5 (5)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 4 (4) | 0 (0)
Lipase increased (Investigations) | 3 (3) | 2 (2)
Liver function test increased (Investigations) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 5 (6)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal vein compression (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Extubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 3 (4)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin Alone (N=975) | Indomethacin+Pancreatic Stent (N=975)
Abdominal pain (Gastrointestinal disorders) | 185 (187) | 188 (189)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 24 (25) | 18 (18)
Vomiting (Gastrointestinal disorders) | 5 (5) | 9 (9)
Pyrexia (General disorders) | 8 (8) | 5 (5)
Lipase increased (Investigations) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 3 (3) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
Potential unmasking events occurred and could have influenced care. Decay in secondary outcome blinding, as unblinded clinician could resume care of patient after 48 h. Adjudicators provided radiographic information when assessing PEP severity, which may have influenced decision making. Unblinded endoscopists made procedural decisions, possibly altered according to study arm. Findings may not be applicable to community endoscopists since all sites were tertiary referral centers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT02476279/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT02476279/SAP_001.pdf